CLINICAL TRIAL: NCT01315730
Title: The Effects of Tactile Speech Feedback on Stuttering Frequency
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Patent being pursued prior to trial initiation
Sponsor: University of Mississippi, Oxford (Other)
Collaborators: West Virginia University (Other); Auburn University (Other); University of Louisiana at Lafayette (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UMO-0001
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Stuttering
Keywords: stuttering; haptic; feedback; fluency
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device: Tactile Stimulation (Experimental): A new medical grade device (FDA - category exempt) has been newly designed and built at the University of Mississippi within the departments of Communication Sciences & Disorders, Exercise Science, and Computer and Electrical Engineering. The device records either sound waves (via a small standard microphone) or three dimensional accelerometer data from the throat of a stuttering subject. This data is digitally signal processed, and "fed back" to the user in the form of a small vibrating disk/film that can be held between the fingers or mounted on the skin. This feedback data does not require the subject to attend to the incoming signal.
  Interventions: Device: Tactile Stimulation

INTERVENTIONS:
Device: Tactile Stimulation — See Arms

SUMMARY:
The purpose of this research project is to test the effects of exposure of different forms of tactile speech feedback on overt stuttering frequency.

DETAILED DESCRIPTION:
A new medical grade device (FDA - category exempt) has been newly designed and built at the University of Mississippi within the departments of Communication Sciences & Disorders, Exercise Science, and Computer and Electrical Engineering. The device records either sound waves (via a small standard microphone) or three dimensional accelerometer data from the throat of a stuttering subject. This data is digitally signal processed, and "fed back" to the user in the form of a small vibrating disk/film that can be held between the fingers or mounted on the skin. This feedback data does not require the subject to attend to the incoming signal.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with persistent developmental stuttering

Exclusion Criteria:

* Subjects below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03

PRIMARY OUTCOMES:
Speech Fluency | 1 week
  Speech fluency was defined by either reading or saying a set syllable sentence in a book which is normally 8th grade reading level or lower. Pauses or stutters are considered positive indicators of dis-fluent speech.

CONTACTS AND LOCATIONS:
Overall Officials: Dwight E Waddell, Ph.D., Principal Investigator — The University of Mississippi
Locations (1):
- The University of Mississippi, University, Mississippi, United States

REFERENCES:
- [Result] Snyder GJ, Blanchet P, Waddell D, Ivy LJ. Effects of digital vibrotactile speech feedback on overt stuttering frequency. Percept Mot Skills. 2009 Feb;108(1):271-80. doi: 10.2466/PMS.108.1.271-280. PMID 19425468